CLINICAL TRIAL: NCT06936605
Title: The Use of Integrin Binding Domain Loaded Hydrogel (RGD) With Minimally Invasive Non-Surgical Technique in Treatment of Periodontal Intrabony Defect (Randomized Clinical Trial Study)
Brief Title: RGD With Minimally Invasive Non-Surgical Technique in Treatment of Periodontal Intrabony Defect
Acronym: MINST + RGD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, lecturer in periodontology, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MINST+ RGD in Periodontitis; committee 1051 (Other: ethical committee faculty of dentistry minia university)
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-01

CONDITIONS: Intrabony Defect; Periodontal Diseases; Alveolar Bone Loss
Keywords: MINST; RGD; intrabony defect
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss | interventions — arginyl-glycyl-aspartic acid

STUDY DESIGN:
Intervention Model Description: Groups and intervention:
  Patients selected in this study will be classified into three groups:
  * Group 1: Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with modified minimally invasive surgical technique (MINST) and RGD hydrogel injection.
  * Group 2: Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with (MINST) and hydrogel injection.
  * Group : Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with (MINST) alone.
  Postoperative phase:
  1. Routine verbal and written postoperative instructions will be given to all patients.
  2. Patients will be advised to refrain from retracting the cheeks, to accomplish food mastication in areas away from surgical site, and to avoid brushing the area in the first week.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients do not know the type of treatment and outcomes assessor does not know type of group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- negative control group (Placebo Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with minimally invasive non-surgical technique
  Interventions: Drug: RGD Peptide
- control group (Placebo Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with minimally invasive non-surgical technique with placebo hydrogel
  Interventions: Drug: RGD Peptide
- study group (Active Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with minimally invasive non-surgical technique with RGD hydrogel
  Interventions: Drug: RGD Peptide

INTERVENTIONS:
Drug: RGD Peptide — RGD peptide is an integrin binding site

SUMMARY:
Periodontal regeneration is a complex process that involves coordinated activities and interactions of many cell types, extracellular matrix, cytokines, and specific growth factors to restore tissue integrity. The most important challenge facing periodontal regeneration is cellular insufficiency. Periodontal defects usually have a limited regenerative capacity due to their bounded surface area which is supposed to provide the wound area with a limited number of viable cells and a limited amount of biologic mediators. Cell recruitment and adhesion into the defect area are essential for cells to survive and secrete collagen.

Apoptosis is initiated when failure in adhesion in many different cell types occurs. Some periodontal treatment options failed in the reconstruction of the defect due to failure in wound stabilization and subsequent cell adhesion. Many treatment options have been developed to enhance defect stability and cellular recruitment including the use of GTM and different biologics. However, the treatment outcomes vary considerably depending on the level of the defect cellularity and the degree of cell recruitment into the defect area. For maximum outcomes, enhanced stability, vascularity, and biologics-sustained delivery were suggested. The minimally invasive surgical technique (MIST) suggested by Cortellini et al. offers a suitable level of tissue preservation that could help in defect stability and cellular adhesion. It was suggested to promote flap stability, maintain space, and maintain a greater amount of blood supply at the alveolar crest and papillary levels.

DETAILED DESCRIPTION:
Periodontitis is an inflammatory multifactorial disease initiated by pathogenic bacteria accumulated as a biofilm on the tooth surface leading to clinical attachment loss (CAL), pocket formation (PD), bleeding on probing (BOP), and bone loss which if neglected may lead to increased tooth mobility and final tooth loss. Pathological tooth mobility may arise from extensive alveolar bone loss, traumatic occlusion, acute periodontal inflammation, and apical tooth displacement. Treating tooth mobility can be a challenging process, particularly for patients with severe periodontitis, including those in stage III or IV, who often experience a range of these symptoms. ue to compromised periodontal support. Therefore, effective treatment not only relies on periodontal therapy but also on occlusal stability and tooth splinting

ELIGIBILITY:
Inclusion Criteria:

* • All patients included will have moderate to advanced periodontitis.

  * Patients included in this study will be free from any systemic diseases according to criteria of Modified Cornell Medical Index(10).
  * Patients who had not undergone any type of regenerative periodontal therapy six months prior to the initial examination.

Exclusion Criteria:

* • Patients with systemic diseases, smokers, pregnant (female).

  * Patients received antibiotics or non-steroidal anti-inflammatory drugs six months before the beginning of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
CAL by millimeters | baseline, 3months and 6 months
  Measure clinical attachment loss pre and after-intervention

IPD SHARING:
Plan to Share IPD: No
after complete study and publishing all data well be available

REFERENCES:
- See also: RGD in treatment of intrabony defect — https://doi.org/10.1590/1678-7757-2023-0263